CLINICAL TRIAL: NCT01597999
Title: Accuracy of Magnetic Resonance Imaging (MRI) in Predicting Aggressiveness of Early Breast Cancer According to Molecular Subtypes Identified by ER PR and HER-2 Status
Brief Title: Benefits of Breast MRI for Predicting of Histopathologic Cell Type of Small Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15262; 578/2533(EC4) (Other: IRB)
Record Dates: First submitted 2011-05-13; First posted 2012-05-15 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Invasive Breast Cancer
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No treatment (Other): Accuracy of magnetic resonance imaging (MRI) in predicting aggressiveness of early breast cancer according to molecular subtypes identified by ER PR and HER-2 status ( Additional benefits of magnetic resonance imaging (MRI) with Gadovist in early breast cancer with poor prognostic features )
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — magnetic resonance imaging (MRI) with Gadovist in early breast cancer with poor prognostic features
  Other Names: Magnetic Resonance Imaging

SUMMARY:
This study examines the additional benefits of magnetic resonance imaging (MRI) with Gadovist in early breast cancer with poor prognostic features.

DETAILED DESCRIPTION:
Dedicated Contrast-enhanced Magnetic Resonance Imaging (DCE-MRI)

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive ductal carcinoma
* Patients undergoing DCE-MRI scan which are assessed according to BI-RADS lexicon
* Breast cancer patients with pathological diagnosed invasive ductal carcinoma with hormonal receptor (ER, PR and HER-2) response
* Patients who have signed on informed consent form Patients will undergo MRI imaging and the physicians will practice according to practice guidelines.

Exclusion Criteria:

* Patients under 18 years old or during pregnancy
* Patients with MRI's contraindications e.g. patients with cardiac pacemaker or are allergic to MRI contrast agent Patients with unstable clinical abnormality and might get unexpected clinical treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
study the benefits of DCE-MRI using Gadovist in prognostic determination of early invasive breast cancer | 1 year
  The benefits of breast tumor diagnosis from DCE-MRI in early invasive breast cancer with poor prognostic features

SECONDARY OUTCOMES:
ascertain the accuracy of pre-operative DCE-MRI in terms of detection and characterization of breast cancer, as compared to tissue biopsy. | 1 year
  The comparision between DCE-MRI radiological features in early invasive breast cancer with poor prognostic features and early invasive breast cancer with good prognostic features To ascertain the accuracy of pre-operative DCE-MRI in terms of detection and charecterization of breast cancer, as compared to tissue biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Pornpim Korpraphong, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand